CLINICAL TRIAL: NCT01787708
Title: Efficacy of Red Light in Vitiligo: A Prospective, Single-Blind Randomized Controlled Trial
Brief Title: Efficacy of Red Light in Vitiligo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02235b
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Vitiligo
Keywords: Vitiligo; red; laser; light
MeSH Terms: conditions — Vitiligo; Erythema | interventions — Red Light

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low intensity red laser (Active Comparator): Patients with a vitiligo patch larger than 25cm2 will be recruited. The target patch will be divided into four quadrants. Two opposite quadrants will be shielded by foil and served as control, the third quadrant will be exposed to low intensity red laser (at 3 J/cm¬2), and the fourth quadrant will be exposed to high intensity red light (at 37 J/cm¬2).
  Treatments will be given twice weekly for 10 weeks. This will be followed by assessments at 4, 8, and 12 weeks post treatment.
  Interventions: Procedure: Red light
- High intensity red light (Active Comparator): Patients with a vitiligo patch larger than 25cm2 will be recruited. The target patch will be divided into four quadrants. Two opposite quadrants will be shielded by foil and served as control, the third quadrant will be exposed to low intensity red laser (at 3 J/cm¬2), and the fourth quadrant will be exposed to high intensity red light (at 37 J/cm¬2).
  Treatments will be given twice weekly for 10 weeks. This will be followed by assessments at 4, 8, and 12 weeks post treatment.
  Interventions: Procedure: Red light
- No treatment1 (covered) (No Intervention): Patients with a vitiligo patch larger than 25cm2 will be recruited. The target patch will be divided into four quadrants. Two opposite quadrants will be shielded by foil and served as control, the third quadrant will be exposed to low intensity red laser (at 3 J/cm¬2), and the fourth quadrant will be exposed to high intensity red light (at 37 J/cm¬2).
  Treatments will be given twice weekly for 10 weeks. This will be followed by assessments at 4, 8, and 12 weeks post treatment.
- No treatment2 (covered) (No Intervention): Patients with a vitiligo patch larger than 25cm2 will be recruited. The target patch will be divided into four quadrants. Two opposite quadrants will be shielded by foil and served as control, the third quadrant will be exposed to low intensity red laser (at 3 J/cm¬2), and the fourth quadrant will be exposed to high intensity red light (at 37 J/cm¬2).
  Treatments will be given twice weekly for 10 weeks. This will be followed by assessments at 4, 8, and 12 weeks post treatment.

INTERVENTIONS:
Procedure: Red light
  Arms: High intensity red light; Low intensity red laser

SUMMARY:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin. There are many treatment modalities available for vitiligo, however, none of them cure the disease. Visible red light has been shown to stimulates melanocyte migration and proliferation resulting in repigmentation of vitiligo patches. However, there are only a few studies published on the efficacy of red light in vitiligo. This is a prospective single-blind randomized clinical trial to assess efficacy of red light in the treatment of vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin and mucous membranes. Mucocutaneous lesions develop secondary to selective destruction of melanocytes. The etiology of vitiligo is largely unknown but more likely to be multifactorial. There are several theories on the pathogenesis of vitiligo including mainly the autoimmune, neurohormonal, and autocytotoxic theories. The autoimmune hypothesis has the strongest evidence with alteration mainly in the cellular immune response.

There are many treatment modalities available for vitiligo, however, none of them cure the disease. These include different topical treatments, phototherapy, surgical therapy, and depigmentation therapy. Visible red light has been shown to stimulates melanocyte migration and proliferation resulting in repigmentation of vitiligo patches. However, there are only a few studies published on the efficacy of red light in vitiligo. The investigators plan on conducting a prospective single-blind randomized clinical trial to assess efficacy of red light in the treatment of vitiligo.

Study Objective To evaluate the potential for red light to induce repigmentation within vitiligo patches.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Localized or generalized vitiligo that involves a non mucosal or acral site.
* Patients should have a patch of at least 25 cm2 that shows no more than 10% repigmentation as assessed visually

Exclusion Criteria:

* Patients who received treatment for vitiligo within the past 3 weeks.
* Patients known to have a photosensitivity disorder
* History of previous skin cancer.
* History of severe medical illness or immunosuppression.
* Pregnancy or breast-feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in the modified VASI score compared to baseline. | assessments at 2, 4, 6, 8 and 10 weeks during treatment then at 4, 8, and 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lui, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, British Columbia, Canada